CLINICAL TRIAL: NCT02949765
Title: Effects of a Dietary Approach to Iron Deficiency in Premenopausal Women Affected by Celiac Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Francesca Ferretti, MD, MD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atto 302/2016
Record Dates: First submitted 2016-09-21; First posted 2016-10-31 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Celiac Disease; Iron Deficiency (Without Anemia)
MeSH Terms: conditions — Celiac Disease; Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron sulfate 105 mg (Active Comparator): Iron sulfate 105 mg: 1 pill/day is administered
  Interventions: Drug: Iron sulfate 105 mg
- Iron-rich diet (Experimental): Iron-rich diet recommendations are given
  Interventions: Dietary Supplement: Iron-rich diet

INTERVENTIONS:
Drug: Iron sulfate 105 mg — Daily supplementation with iron sulfate 105 mg 1 pill/day
  Arms: Iron sulfate 105 mg
Dietary Supplement: Iron-rich diet
  Arms: Iron-rich diet

SUMMARY:
Anemia and sideropenia are a common effect of untreated celiac disease. In a portion of patients a certain degree of hypoferritinemia persist after the diagnosis, despite a good compliance and clinical response to gluten-free diet. These patients are usually premenopausal women in whom the cyclic menstrual bleeding and the oral iron intake are not balanced.

The aim of the study is to compare the efficacy of a pharmacological therapy, frequently not tolerated, and a dietary approach through a iron-rich diet in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Celiac patients on gluten free diet since 1 year
* iron deficiency (ferritin <15 ng/L or ferritin 15-20 + transferrin saturation <15%)

Exclusion Criteria:

* allergy to iron supplementation
* anemia
* pregnancy or breastfeeding
* menopause
* organic or psychiatric diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Ferritin levels (ng/mL) increase > 95% compared to basal levels | 12 weeks

SECONDARY OUTCOMES:
Hemoglobin levels (g/dL), compared to basal levels | 12 weeks
Iron levels (mcd/dl), compared to basal levels | 12 weeks
Transferrin saturation (%, ratio of serum iron and total iron-binding capacity), compared to basal levels | 12 weeks

OTHER OUTCOMES:
Number of participants with treatment-related adverse events assessed through NRS (number rating scales) | 12 weeks
Degree of compliance to therapy assessed through telephone interviews (number of pills taken) | 12 weeks
Degree of compliance to diet assessed through compliance questionnaires (mg of irons ingested) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Francesca, MD, Principal Investigator — Gastroenterology and Endoscopy Unit Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico Department of Pathophysiology and Transplantation Università degli Studi di Milano - Italy.
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No